CLINICAL TRIAL: NCT05498285
Title: A Pilot Single-blind Parallel Randomised Controlled Trial Comparing Mobile App (UPSCALER) to Standard Care in the Rehabilitation of ACL Injury After Reconstructive Surgery
Brief Title: Post-ACL Reconstruction Rehab UPSCALER App RCT HPUPM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Pengajar Universiti Putra Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JKEUPM-2022-294
Record Dates: First submitted 2022-08-08; First posted 2022-08-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: ACL Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Use of UPSCALER App
  Interventions: Behavioral: UPSCALER app
- Control (No Intervention): No app used. Conventional treatment.

INTERVENTIONS:
Behavioral: UPSCALER app — Usage of mobile app to guide rehabilitation after surgery
  Arms: Intervention

SUMMARY:
EXECUTIVE SUMMARY

Research Title An Android Application-Based Delivery of Guided Rehabilitation After Anterior Cruciate Ligament Reconstruction: A Randomised Single-Blinded Pilot Study

Investigators Principle Investigator (Supervisor) : Prof Madya Dr Mohd Nizlan Mohd Nasir Co-investigator (Supervisor) : Dr Khairil Anwar bin Ahmad Hanif Dr Firdati binti Mohamed Saaid Co-Investigator (Student) : Dr Tan Eng Kee

Background Anterior cruciate ligament injuries are a common and significant injury seen in active persons. This injury can adversely affect the patient's daily life, as well as delay or prevent return to sports, in addition to predisposing patients to long-tern knee conditions such as osteoarthritis. Despite surgical advances, ACL reconstruction surgery outcomes are still considered poor, with a low as 55% of patients returning to active sports. One of the key factors that lead to a poorer outcome is the patient's compliance to rehabilitation, causing less than satisfactory results in the post-operative period. With the conventional regime, rehabilitation typically takes one year. Patients tend to drop out of the rehabilitation regime due to its long duration. In order to combat this, the accelerated regime was developed and only took 6 months. This regime has been researched and validated by numerous international publications since its inception. However, compliance remained poor.

Purpose of Study The study aims to assess the feasibility and effectiveness of a smartphone-based application to guide the patient's rehabilitation regime and improve compliance.

Data Gathering and Analysis Data for outcome assessment will be obtained via a patient administered questionnaire called the Knee Injury and Osteoarthritis Outcome Score (KOOS). This scoring system is available for free without licensing requirements, and has been validated by numerous research publications internationally.

Analysis of obtained data will be performed using SPSS version 22. Continuous data will be displayed as mean + SD as well as median.

Conclusion There is a need for a new method of information provision as the country moves towards the age of information technology. This smartphone-based application for guided rehabilitation will be an innovative new method to aid patients.

Lastly, the researchers would like to thank the members of JKEUPM for their time, effort and kind consideration of this research proposal.

DETAILED DESCRIPTION:
Study Design:

Single-blinded randomized control pilot study

Study Location:

Hospital Pengajar Universiti Putra Malaysia Orthopaedic Department

Study Duration:

1 year (September 2022 to August 2023)

Study Population:

Consenting patients from HPUPM Orthopaedic Department, SIASCOE Unit who are undergo elective arthroscopic ACL reconstruction surgery

Sample Size:

The sample size for this study was concluded to be 30 based on the objectives. Different sample sizes were calculated and the highest number was taken. (See Appendix A)

Patient Recruitment:

Patients from the SIASCOE clinic who fall within the inclusion criteria will be informed regarding this research using the patient's information sheet. Should they choose to join the research; consent will be obtained with a witness present.

They will also be informed as any patient would, that the surgery will be performed by the same team using the anatomical ACL reconstruction technique. Concomitant procedures such as meniscectomy or meniscal repair, operative time as well as tourniquet time and pressure will be recorded as with any other patient who undergoes an ACL reconstruction. Post-operative precautions will be taken as with any patient. A hinge knee brace and a compressive wrap will be used immediately post-op, cryocuff therapy started once patient is back in the ward.

Patient Randomization Patients will be randomized into treatment or control arm based on the last digit of their UPM registration number. Even numbers for treatment, and odd numbers for control.Patient forms will be colour coded to either red or blue for blinding of the researcher. Patients in the control arm will not be informed of the usage of the app as it may create a bias.

Data Collection and Researcher Blinding KOOS forms will be provided to the participant. They will be placed in a private setting during the self-administered assessment with an investigator available for any queries. Privacy and confidentiality will be ensured and there will be no personal data included in the KOOS forms. All participants will be assigned an identification number known only to the primary researcher and all KOOS forms will be colour coded to indicate the randomly assigned group of the participant.

SIRAS assessment forms will also be provided to patients during follow up to assess adherence to the rehabilitation regime. This assessment form will be filled by the physician and consist of three items that assess the patient's intensity during rehabilitation, ability to follow instructions, and their receptiveness to the rehabilitation.

Two researchers will be allocated for data collection. Researcher A will obtain data related to KOOS and SIRAS scoring. This researcher will be blinded and provided with colour coded forms according to the group that the patient has been randomized to.

Researcher B will obtain data related to acceptance of the mobile app. This researcher is unable to be blinded and will only be allocated to patients in the treatment group.

The data collected by this Researcher B will be stored in a separate location from the data collected by Researcher A until the study is completed. They will only be compiled immediately prior to data analysis.

ELIGIBILITY:
Inclusion criteria:

* Male and female
* Patients above the age of 18
* Patients with ACL injury who undergo ACL reconstruction surgery with or without meniscectomy
* Patients who receive autologous hamstring grafts for ACL reconstruction
* Malaysian

Exclusion criteria:

* Patients below the age of 18
* Patients unwilling to participate
* Patients with concurrent injuries to other structures in the ipsilateral knee e.g. multiligamentous injuries
* Non-Malaysian
* Patients who require meniscus repair instead of meniscectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
KOOS score | 6 months
  Pattient administered scoring system

CONTACTS AND LOCATIONS:
Overall Officials: Eng Kee Tan, MBBS, Principal Investigator — Hospital Pengajar Universiti Putra Malaysia
Locations (1):
- Hospital Pengajar Universiti Putra Malaysia, Serdang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No